CLINICAL TRIAL: NCT06345105
Title: Prospective Evalulation of Artificial Intelligence-assisted Monitoring of Effective Withdrawal Time Versus Standard Withdrawal Time on Adenoma Detected Per Colonoscopy
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: AIeffectiveV4
Record Dates: First submitted 2024-03-22; First posted 2024-04-03 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2023-11

CONDITIONS: Colon Polyp; Colon Adenoma; Artificial Intelligence
Keywords: Colon Polyp; Artificial Intelligence; Withdrawal time
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AI group: AI monitoring of effective withdrawal time
  Interventions: Device: Endoscreener QC

INTERVENTIONS:
Device: Endoscreener QC — Artificial intelligence monitoring of effective withdrawal time

SUMMARY:
The goal of this observational study is to assess the correlation between the artificial intelligence (AI) derived effective withdrawal time (EWT) during colonoscopy and endoscopists' adenoma per colonoscopy (APC), polyp per colonoscopy(PPC), adenoma detection rate (ADR), polyp detection rate (PDR) and during colonoscopy for each endoscopists. The association between the AI derived EWT with all colonoscopy outcomes during the prospective colonoscopy series would also be determined. The colonoscopy video of participants will be monitored by the AI. The result will be compared with standard withdrawal time (SWT).

DETAILED DESCRIPTION:
This is a prospective colonoscopy trial using artificial intelligence (AI) real time effective mucosal examination monitor system (EndoScreener QC, Wision A.I. Shanghai & Chengdu). Low residue diet will be taken by all patients two days before the scheduled colonoscopy. Oral polyethylene glycol lavage solution is used for bowel preparation as in usual hospital practice. All examination will be performed with high-definition endoscopes (EVIS-EXERA 290 video system, Olympus Optical, Tokyo, Japan) under white light by experienced endoscopists. In all colonoscopy examination, colonoscope will be first advanced to the cecum as confirmed by identification of the appendiceal orifice and ileocecal valve or by intubation of the ileum. After cecal intubation is performed, the colonoscopy is slowly withdrawn. All detected polyps will be removed during the withdrawal only. The size (measured with biopsy forceps), location and morphology of each polyp will be recorded by an independent observer. The withdrawal time (minus the polypectomy site) will be measured by a stopwatch and with a minimum of 6 minutes. The bowel preparation quality will be graded according to the Boston Bowel Preparation Scale. The AI derived (AI) real time effective mucosal examination monitor system (EndoScreen QC) will be initiated during scope withdrawal, starting from cecum to anus. The polypectomy or biopsy time will be removed as determination of standard withdrawal time. All endoscopists will be blinded to the results of AI real time monitoring of EWT. All polyp specimens removed will be clearly labelled and send for histological examination. All resected and biopsy specimens are fixed in 10% buffered formalin solution, and examined histologically by hematoxylin and eosin staining. The histopathological diagnosis is determined by experienced pathologists, who are blinded to the assigned endoscopic system, according to the World Health Organization (WHO) criteria. Advanced adenomas are defined as adenoma ≥10 mm in diameter or with villous histology in 25% or high-grade dysplasia (HGD), or carcinoma.The primary outcome of this study is to correlate the adenoma detection rates of the endoscopists with EWT.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients, aged 40 or above, undergoing outpatient colonoscopy will be recruited

Exclusion Criteria:

* history of inflammatory bowel disease
* history of colorectal cancer
* previous bowel resection (apart from appendectomy)
* Peutz-Jeghers syndrome, familial adenomatous polyposis or other polyposis syndromes
* bleeding tendency or severe comorbid illnesses for which polypectomy is considered unsafe.
* Cecum could not be intubated for various reasons
* Poor bowel preparation with Boston Bowel Preparation Scale (BBPS) < 6

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patient will be recruited in Queen Mary Hospital, Hong Kong, China
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Adenoma per colonoscopy of the endoscopists | During the colonoscopy
  Adenoma per colonoscopy of the endoscopists

SECONDARY OUTCOMES:
Adenoma detection rate of the endoscopists | During that colonoscopy
  Adenoma detection rate of the endoscopists
Polyp detection rate of the endoscopists | During that colonoscopy
  Polyp detection rate of the endoscopists
Polyp per colonoscopy of the endoscopists | During colonoscopy
  Polyp per colonoscopy of the endoscopists
Serrated Lesion per Colonoscopy of the endoscopist | During the colonoscopy
  Serrated Lesion per Colonoscopy of the endoscopist
Serrated Lesion Detection Rate of the endoscopist | During colonoscopy
  Serrated Lesion Detection Rate of the endoscopist

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ka-Luen Lui, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, the University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided